CLINICAL TRIAL: NCT00002343
Title: An Open-Label Randomized Pharmacokinetic/Pharmacodynamic Study of Mycobutin (Rifabutin) or Rifabutin in Combination With Myambutol (Ethambutol) for Prophylaxis of Mycobacterium Avium Complex (MAC) Bacteremia in AIDS Patients With CD4 Counts <= 100 Cells/mm3
Brief Title: A Study of Rifabutin, Used Alone or With Ethambutol in the Prevention of Mycobacterium Avium Complex (MAC) Bacteremia in Patients With AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 048E; CS 087287-000
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-06

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Rifabutin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Rifabutin

SUMMARY:
To optimize Mycobacterium avium Complex (MAC) prophylaxis in AIDS patients by measuring serum rifabutin levels and adjusting the dose accordingly. To combine rifabutin with ethambutol to examine the effect of combination therapy in preventing or delaying the incidence of MAC bacteremia in this patient population.

DETAILED DESCRIPTION:
Patients are randomized to receive oral rifabutin alone or rifabutin/ethambutol daily for 12 months, with possible continuation of medicine lifelong. Doses will be adjusted to maintain minimum blood levels of the drugs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* AZT, d4T, ddI, or ddC.
* Antipneumocystis prophylaxis.

Allowed:

* Short course (< 14 days) of ciprofloxacin for acute infections.

Patients must have:

* AIDS.
* CD4 count <= 100 cells/mm3.
* NO prior or current MAC infection.

Prior Medication:

Required:

* Antipneumocystis prophylaxis for at least 4 weeks prior to study entry.

Allowed:

* Prior rifabutin.
* Prior ethambutol.
* Prior clarithromycin.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Positive tuberculin skin test (PPD > 5 mm).
* Active M. tuberculosis.
* Perceived as unreliable or unavailable for frequent monitoring.

Concurrent Medication:

Excluded:

* Other antiretrovirals not specifically allowed.
* All investigational drugs.
* Other antimycobacterial therapy, such as clarithromycin, azithromycin, rifampin, clofazimine, amikacin, streptomycin, isoniazid, cycloserine, ethionamide, and ciprofloxacin (>= 14 days).

Patients with the following prior conditions are excluded:

Known hypersensitivity to rifabutin, rifampin, or other rifamycins and/or ethambutol.

Prior Medication:

Excluded within 4 weeks prior to study entry:

* Rifampin.
* Isoniazid.
* Clofazimine.
* Cycloserine.
* Ethionamide.
* Amikacin.
* Ciprofloxacin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of California - Davis Med Ctr / CARES, Sacramento, California, United States